CLINICAL TRIAL: NCT02115451
Title: Dynamic Stability of the ACL Deficient Knee
Brief Title: Nonsurgical or Surgical Treatment of ACL Injuries
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Other Study IDs: 685-06289
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical treatment: Patients who undergo rehabilitation and anterior cruciate ligament reconstruction, other surgical interventions may be performed
- Nonsurgical treatment: Patients who undergo rehabilitation without anterior cruciate ligament reconstruction, other surgical interventions may be performed

SUMMARY:
The aim of this study is to evaluate knee function, sports participation and knee reinjuries over 2 years in a group of patients who choose either nonsurgical or surgical treatment for an anterior cruciate ligament (ACL) injury

DETAILED DESCRIPTION:
This study is a part study of an overall study with the title 'Dynamic stability of the ACL-injured knee'. The overall study prospectively follows a cohort of newly injured patients with total rupture of the anterior cruciate ligament in the knee.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament rupture within 3 months of injury
* Preinjury participation in level I or II sports at least twice a week

Exclusion Criteria:

* Current or previous injury to the contralateral leg
* Another grade III ligament injury, fracture, full-thickness articular cartilage damage

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Athletically active anterior cruciate ligament injured patients
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2007-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Patient-reported knee function (IKDC 2000) | 2 years

SECONDARY OUTCOMES:
Isokinetic knee extensor and flexor muscle strength | 2 years
Knee reinjury | 2 years
Participation in level I, II and III sports | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT PhD, Principal Investigator — Norwegian Research Center for Active Rehabilitation
Locations (1):
- NAR- Department of Orthopaedics, Oslo University Hospital & Nimi, Oslo, Oslo County, Norway